CLINICAL TRIAL: NCT02040597
Title: Open-label, Non-randomized, Parallel-group Study to Investigate the Pharmacokinetics, Safety and Tolerability of a Single Dose of CHF 5993 pMDI in Subjects With Mild, Moderate and Severe Renal Impairment in Comparison With Matched Healthy Control Subjects.
Brief Title: A Study to Investigate the Pharmacokinetics, Safety and Tolerability of CHF 5993 pMDI in Subjects With Renal Impairment.
Acronym: TRIPLE10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCD-05993AA1-10; 2013-002140-91 (EudraCT Number)
Record Dates: First submitted 2014-01-09; First posted 2014-01-20 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHF5993 pMDI (Experimental): CHF 5993 pMDI (Beclometasone/Formoterol/Glycopyrrolate 100/6/25 mcg) 4 inhalations
  Interventions: Drug: Beclometasone/Formoterol/Glycopyrrolate

INTERVENTIONS:
Drug: Beclometasone/Formoterol/Glycopyrrolate
  Other Names: CHF 5993 pMDI

SUMMARY:
The study is performed to characterize the pharmacokinetics of glycopyrrolate bromide after single administration of CHF 5993 pressurised Metered Dose Inhaler (pMDI) in subjects with different level of renal impairment in comparison with matching healthy volunteers. Moreover, the safety and tolerability of the study drug will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and
* Subjects with mild, moderate and severe renal impairment

Exclusion Criteria:

* pregnant or lactating women
* positive HIV and hepatitis serology
* history of drug abuse
* history of hypersensitivity to the products used in the trial
* smokers
* respiratory disease such as asthma and COPD
* clinically relevant concomitant disease that may introduce a risk for the subjects'safety
* presence of kidney stones
* dialysis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Glycopyrrolate area under the curve (AUC) | over 72 h after single administration
  AUC until the last quantifiable concentration (AUCt)

SECONDARY OUTCOMES:
Glycopyrrolate other Pharmacokinetic parameters in plasma | Over 72 h after single administration
  AUC until 72 h post dose (AUC0-72h), AUC extrapolated to infinity (AUCinf), maximum plasma concentratio (Cmax), time to maximum plasma concentration (tmax), half-life, clearance
B17MP and Formoterol pharmacokinetic parameters in plasma | over 24 h after single administration
  AUCt, AUC until 24 h post dose (AUC0-24h), AUCinf, Cmax, tmax, half-life, clearance
BDP pharmacokinetic parameters in plasma | over 24 h after single administration
  AUCt, AUCinf, Cmax, tmax, half-life
Urine Glycopyrrolate excretion (Ae) | over 72 h after single administration
Urine formoterol excretion (Ae) | Over 24 h after single administration
Adverse events | A period of 3 to 7 weeks (from screening visit to follow-up phone call)
  This includes a period of 3 to 7 weeks (depending on duration of screening and follow-up periods), before and after the study drug administration
Vital signs | over 24 h after single administration
  systolic and diastolic blood pressure
Electrocardiogram (ECG) parameters | over 24 h after single administration
  Heart rate (HR), time interval between ECG waves Q and T corrected for heart rate with Fridericia's formula (QTcF), time interval between the onset of the ECG wave P and the start of the QRS complex (PR), time interval between the beginning of Q wave and the termination of the S wave (QRS)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, MD, Principal Investigator — Medical University in Lodz; Kasia Jarus-Dziedzic, MD, Principal Investigator — Biovirtus
Locations (2):
- Poland (2):
  - Biovirtus Research Site, Nadarzyn, Mokra 7
  - Medical University in Lodz, Lodz, Ul. Kopcińskiego 22

REFERENCES:
- See also: CSR Synopsis available in the Chiesi Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-05993AA1-10.pdf